CLINICAL TRIAL: NCT01252433
Title: Children's Intake of Foods Reduced in Energy Density
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Barbara J. Rolls, Professor of Nutrition and Director of the Laboratory for the Study of Human Ingestive Behavior, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: FoodED201; R01DK082580 (NIH)
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Vegetable Intake

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Entree energy density 100% (Experimental): 100% energy density
  Interventions: Other: Energy density feeding study
- Entree energy density 85% (Experimental): 85% energy density
  Interventions: Other: Energy density feeding study
- Entree energy density 75% (Experimental): 75% energy density
  Interventions: Other: Energy density feeding study

INTERVENTIONS:
Other: Energy density feeding study — In a crossover study, children are served all foods 1 day a week for 3 weeks. Meal entrees will vary in energy density (100%, 85%, 75%).

SUMMARY:
The purpose of this research is to investigate children's responses to incorporating vegetables into selected entrees and snacks over several days. The hypothesis is that children will increase their vegetable intake by consuming foods that have been reduced in energy density through the addition of vegetables. Effects on energy intake will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* enrolled in daycare centers at Penn State University

Exclusion Criteria:

* food allergies or intolerances

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2010-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Food intake | 1 month

SECONDARY OUTCOMES:
Energy intake | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

REFERENCES:
- [Derived] Spill MK, Birch LL, Roe LS, Rolls BJ. Hiding vegetables to reduce energy density: an effective strategy to increase children's vegetable intake and reduce energy intake. Am J Clin Nutr. 2011 Sep;94(3):735-41. doi: 10.3945/ajcn.111.015206. Epub 2011 Jul 20. PMID 21775554